CLINICAL TRIAL: NCT07295574
Title: Digital Occlusal Analysis and Bite Force Evaluation of Hall Technique Vs Stainless-Steel Crowns as Conventional Restoration of Carious Primary Molars Using T-scan: A Randomized Clinical Trial
Brief Title: Digital Occlusal Analysis and Bite Force Evaluation of the Hall Technique Vs Stainless Steel Crowns in Primary Molars Using T-scan
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lujain Yasser Wagih Youssef, Master's Student, Department of Pediatric Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HT-SSC-TSCAN-RCT-2025
Record Dates: First submitted 2025-12-03; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Carious Primary Molars; Bite Force; Occlusal Analysis; Stainless-steel Crown
Keywords: Hall Technique; Stainless Steel Crown; Carious Primary Molars; Digital Occlusal Analysis; T-Scan; Bite Force; Occlusal Force Distribution; Vertical Dimension; Pediatric Dentistry; Minimal Intervention Dentistry; Conventional Crown Preparation; Randomized Clinical Trial

STUDY DESIGN:
Intervention Model Description: This study is designed as a prospective, parallel group, randomized controlled clinical trial with a 1:1 allocation ratio, comparing two restorative techniques for carious primary molars: the Hall Technique (intervention) and the conventional stainless-steel crown (control).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hall Technique Stainless-Steel Crown Placement (Experimental): Participants in this arm will receive a stainless-steel crown (NuSmile) placed using the Hall Technique, a minimally invasive method that does not require local anesthesia, caries removal, or tooth preparation. The appropriately sized crown will be selected based on mesiodistal measurements and trial fitting, then cemented using glass ionomer luting cement. Orthodontic separators may be placed when contacts are tight. Outcome measurements (T-Scan bite force, vertical dimension, questionnaires) will be taken at baseline, immediately after placement, and at 2- and 4-week follow-ups.
  Interventions: Procedure: Hall Technique Stainless Steel Crown Placement
- Conventional Stainless-Steel Crown Restoration (Active Comparator): Participants in this arm will receive a stainless-steel crown (NuSmile) placed using the traditional conventional technique. This includes local anesthesia, complete caries removal, and tooth preparation (occlusal reduction ~1.5 mm, proximal slicing). The crown will be fitted, adjusted for proper occlusion, and cemented using glass ionomer luting cement. Standardized outcome measurements (T-Scan bite force, vertical dimension, questionnaires) will be recorded at baseline, immediately post-operatively, and at 2- and 4-week follow-ups.
  Interventions: Procedure: Conventional Stainless Steel Crown Placement

INTERVENTIONS:
Procedure: Hall Technique Stainless Steel Crown Placement — Children allocated to the intervention group will receive stainless-steel crown (SSC) placement using the Hall technique, without local anesthesia, caries removal, or tooth preparation. An appropriately sized preformed stainless-steel crown (NuSmile®) will be selected based on mesiodistal width and crown fit, and cemented using glass ionomer luting cement. Orthodontic separators may be placed when required to facilitate crown seating. No occlusal adjustment will be performed. Digital occlusal analysis and bite force assessment will be conducted using the T-Scan system, and vertical dimension will be measured using a digital caliper preoperatively, immediately after crown placement, and during the follow-up period according to the study schedule.
  Arms: Hall Technique Stainless-Steel Crown Placement
Procedure: Conventional Stainless Steel Crown Placement — Children allocated to the control group will receive conventional stainless-steel crown (SSC) restoration under local anesthesia following complete caries removal and standard tooth preparation, including occlusal reduction and proximal slicing. An appropriately sized preformed stainless-steel crown (NuSmile®) will be selected, adjusted if necessary, and cemented using glass ionomer luting cement. Occlusion will be clinically adjusted to eliminate premature contacts. Digital occlusal analysis and bite force assessment will be performed using the T-Scan system, and vertical dimension will be measured using a digital caliper preoperatively, immediately after crown placement, and during the follow-up period according to the study schedule.
  Arms: Conventional Stainless-Steel Crown Restoration

SUMMARY:
This randomized controlled clinical trial aims to compare two restorative techniques for managing carious primary molars in children aged 6-9 years: the Hall Technique and conventional stainless-steel crown (SSC) placement. The study evaluates how each technique affects occlusal force distribution, mean bite force, and vertical dimension changes using the T-Scan digital occlusal analysis system. Additional outcomes include temporomandibular joint assessment, child discomfort levels, and parental satisfaction with treatment. Participants are allocated 1:1 to receive either the Hall Technique or conventional SSC restoration, and outcomes are measured at baseline, immediately after treatment, and at 2- and 4-week follow-ups. The study aims to determine whether the minimally invasive Hall Technique provides comparable occlusal function and patient-centered outcomes when compared to traditional SSC preparation methods.

DETAILED DESCRIPTION:
This randomized controlled clinical trial evaluates the effect of two restorative techniques-the Hall Technique and conventional stainless-steel crown (SSC) placement-on digital occlusal parameters and bite force distribution in carious primary molars. The study uses T-Scan digital occlusal analysis to objectively measure changes in occlusion and vertical dimension following restoration.

Children aged 6-9 years presenting with symptomless carious primary molars without pulpal involvement are eligible for inclusion. Participants are randomly assigned (1:1) to receive either an SSC placed using the Hall Technique (no caries removal or tooth preparation) or an SSC placed using the conventional technique (local anesthesia, caries removal, and tooth preparation). All clinical procedures are performed by a single operator to minimize performance bias, and the statistician is blinded during data analysis.

Digital occlusal analysis is conducted using T-Scan Novus to measure bite force percentage and maximum intercuspal position at baseline, immediately after crown placement, and at follow-up visits (2 and 4 weeks). Changes in vertical dimension are evaluated using a digital caliper at the same intervals. Secondary assessments include temporomandibular signs and symptoms, child discomfort, and parental satisfaction using validated questionnaires.

The primary objective is to compare mean biting force between the two restorative techniques over time. Secondary outcomes include changes in vertical dimension, presence of TMD-related symptoms, and subjective evaluations of comfort and esthetics. The study aims to provide clinical evidence regarding differences in occlusal equilibration and functional adaptation between biological minimally invasive management (Hall Technique) and the conventional restorative approach for carious primary molars.

Results from this trial may help guide clinical decision-making regarding restorative methods that optimize occlusion, patient comfort, and treatment acceptance in pediatric dentistry.

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy children
2. Age ranging from 6 to 9 years
3. Cooperative behavior (positive rating on the Frankl Behavior Rating Scale)
4. Unrestored carious primary molar
5. Extent of caries radiographically confined to dentin (≤ or > ½ dentin thickness)
6. Tooth must be vital and symptomless, with no clinical or radiographic signs of pulpal pathology

Exclusion Criteria:

1. Children with special health care needs
2. Temporomandibular disorders, bruxism or parafunctional habits
3. pathological facial swelling
4. periodontal diseases such as gingivitis, drug-induced gingival enlargement, juvenile or aggressive periodontitis
5. Any child showing mobility, bone loss, or signs of pulpal pathology is also excluded from the study.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Mean Bite Force | Baseline (pre-operative), immediate post-operative, 2 weeks post-operative, 4 weeks post-operative
  Occlusal evaluation for bite force will be done using T-Scan III. Changes in bite force at different periods will be assessed using a standardized T-Scan III Software. The obtained bite force will be recorded in percentage concerning the crowned tooth, opposing tooth, right and left side of the arch, during preoperative, postoperative and follow up periods after 2 and 4 weeks. The maximum intercuspal position (MIP) will be measured by changes in the bite force %.

SECONDARY OUTCOMES:
Change in Vertical Dimension | Baseline (pre-operative), immediate post-operative, 2 weeks post-operative, 4 weeks post-operative
  The vertical dimension will be assessed to evaluate any changes in occlusal height following crown placement using either the Hall technique or the conventional stainless steel crown technique. Measurements will be taken using a digital caliper at four time points: preoperatively, immediately after crown placement, at 2 weeks, and at 4 weeks postoperatively. The vertical distance of the overbite will be measured in millimeters between the maxillary and mandibular canines while the child is in maximum intercuspal position. This outcome is used to detect temporary occlusal discrepancies and to monitor the process of occlusal re-equilibration over time following crown placement.
Temporomandibular Joint (TMJ) Assessment | Baseline (pre-operative) and 4 weeks post-operative
  Temporomandibular joint status will be evaluated using a standardized questionnaire based on the American Academy of Pediatric Dentistry (AAPD) guidelines. The assessment consists of binary (yes/no) questions addressing symptoms such as pain during chewing, jaw clicking, difficulty in mouth opening, jaw locking, or discomfort around the ears and cheeks. This outcome is measured to detect any functional disturbance associated with changes in occlusion after stainless steel crown placement by either technique.
Child Discomfort Level | Immediate post-operative and 4 weeks post-operative
  The level of discomfort experienced by the child after crown placement will be assessed using the Wong-Baker FACES Pain Rating Scale. This validated tool allows children to express their perceived pain using facial expressions representing increasing levels of discomfort, ranging from 0 (no pain, smiling face) to 10 (worst pain, crying face), with intermediate scores of 2, 4, 6, and 8 corresponding to increasing pain intensity. This outcome helps compare patient tolerance and comfort between the minimally invasive Hall technique and the conventional stainless ste
Parental Satisfaction with Esthetics | Immediate post-operative and 4 weeks post-operative
  Parental satisfaction with the esthetic appearance of the crown will be assessed using a structured questionnaire based on a five-point Likert scale. Parents will be asked to rate the size, shape, color, and overall appearance of the crown, with responses ranging from 1 (very dissatisfied), 2 (dissatisfied), 3 (neutral), 4 (satisfied), to 5 (very satisfied).
Parental Perception of Treatment Impact on the Child | Immediate post-operative and 4 weeks post-operative
  Parents will evaluate the overall impact of the treatment on their child using a structured questionnaire with a five-point Likert scale, with responses ranging from 1 (not at all satisfied) to 5 (very much satisfied). The questionnaire will assess the following aspects: improvement in the child's oral health after crown placement, parents' concern about the appearance of the teeth before crowns, whether the child avoided smiling before crowns, whether the child smiled after crowns, and whether the crowns improved the overall appearance of the child's teeth. This outcome helps assess the psychosocial and functional impact of both the Hall technique and the conventional stainless steel crown technique from the caregiver's perspective.

CONTACTS AND LOCATIONS:
Overall Officials: Osama A El Shahawy, PhD, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Umapathy Thimmegowda and Radhakrishnan, A. (2023). Application of Tekscan in Pediatric Dentistry:AReview.pp.132-142. doi:Hall techniquetps://doi.org/10.9734/bpi/cidhr/v1/6603a
- [Background] Schuler IM, Hiller M, Roloff T, Kuhnisch J, Heinrich-Weltzien R. Clinical success of stainless steel crowns placed under general anaesthesia in primary molars: an observational follow up study. J Dent. 2014 Nov;42(11):1396-403. doi: 10.1016/j.jdent.2014.06.009. Epub 2014 Jun 30. PMID 24994618
- [Background] Herkar PP, Anantharaj A, Praveen P, Shankarappa PR, Sudhir R. A comparative study of conventional and Hall techniques of crown placement using finite element stress analysis. J Indian Soc Pedod Prev Dent. 2022 Jul-Sep;40(3):302-310. doi: 10.4103/jisppd.jisppd_173_22. PMID 36260472
- [Background] Rahate I, Fulzele P, Thosar N. Comparative evaluation of clinical performance, child and parental satisfaction of Bioflx, zirconia and stainless steel crowns in pediatric patients. F1000Res. 2023 Dec 21;12:756. doi: 10.12688/f1000research.133464.2. eCollection 2023. PMID 38911945
- [Background] Hu S, BaniHani A, Nevitt S, Maden M, Santamaria RM, Albadri S. Hall technique for primary teeth: A systematic review and meta-analysis. Jpn Dent Sci Rev. 2022 Nov;58:286-297. doi: 10.1016/j.jdsr.2022.09.003. Epub 2022 Sep 27. PMID 36185501
- [Background] Boyd DH, Thomson WM, Leon de la Barra S, Fuge KN, van den Heever R, Butler BM, Leov F, Foster Page LA. A Primary Care Randomized Controlled Trial of Hall and Conventional Restorative Techniques. JDR Clin Trans Res. 2021 Apr;6(2):205-212. doi: 10.1177/2380084420933154. Epub 2020 Jun 19. PMID 32559403
- [Background] Ayedun OS, Oredugba FA, Sote EO. Comparison of the treatment outcomes of the conventional stainless steel crown restorations and the hall technique in the treatment of carious primary molars. Niger J Clin Pract. 2021 Apr;24(4):584-594. doi: 10.4103/njcp.njcp_460_20. PMID 33851682
- [Background] Araujo MP, Uribe S, Robertson MD, Mendes FM, Raggio DP, Innes NPT. The Hall Technique and exfoliation of primary teeth: a retrospective cohort study. Br Dent J. 2020 Feb;228(3):213-217. doi: 10.1038/s41415-020-1251-1. PMID 32060464
- [Background] Amlani DV, Brizuela M. Stainless Steel Crowns in Primary Dentition. 2023 Mar 19. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK574547/ PMID 34662061
- [Result] Nair K, Chikkanarasaiah N, Poovani S, Thumati P. Digital occlusal analysis of vertical dimension and maximum intercuspal position after placement of stainless steel crown using hall technique in children. Int J Paediatr Dent. 2020 Nov;30(6):805-815. doi: 10.1111/ipd.12647. Epub 2020 May 7. PMID 32248585
- [Result] Maheshkumar K, Chowdhary N, Chowdharry R, Vundela RR, Sonnahalli NK, Anuraaga AT. Bite force evaluation at maximal intercuspal position: An in vivo comparative study between stainless steel and zirconia crowns on primary molar teeth. J Indian Soc Pedod Prev Dent. 2023 Apr-Jun;41(2):89-97. doi: 10.4103/jisppd.jisppd_156_23. PMID 37635466
- [Result] Bhatia HP, Khari PM, Sood S, Sharma N, Singh A. Evaluation of Clinical Effectiveness and Patient Acceptance of Hall Technique for Managing Carious Primary Molars: An In Vivo Study. Int J Clin Pediatr Dent. 2019 Nov-Dec;12(6):548-552. doi: 10.5005/jp-journals-10005-1699. PMID 32440073
- [Result] Aishwarya N, Nagarathna C, Poovani S, Thumati P. Comparison of Bite Force and the Influencing Factors Pre- and Post-cementation of Stainless Steel Crown in Children Using T-Scan. Int J Clin Pediatr Dent. 2021 Jan-Feb;14(1):46-50. doi: 10.5005/jp-journals-10005-1900. PMID 34326583